CLINICAL TRIAL: NCT05070299
Title: Developing a Psychosexual Educational Partners Program: PEPP A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: The Breast Cancer Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2021.071; HUM00202063 (Other: University of Michigan)
Record Dates: First submitted 2021-09-21; First posted 2021-10-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosexual Educational Partners Program (PEPP) (Experimental): Women and their partners will work through a three module workbook together, completing each module over a 2-week period (6 weeks total).
  Interventions: Behavioral: Psychosexual Educational Partner Program (PEPP)

INTERVENTIONS:
Behavioral: Psychosexual Educational Partner Program (PEPP) — A communication and intimacy promotion kit consisting of three modules devoted to information sharing, partner communication and activities for building intimacy.

SUMMARY:
This is a single arm study to evaluate the feasibility, adherence, and usefulness of a psychosexual education partner program (PEPP) to improve partner communication and sexual function. This study is intended to get initial input from a small group of up to 10 women and their partners about the appropriateness, usefulness, and critical nature of the content as well as the feasibility and appeal of the method of delivery.

DETAILED DESCRIPTION:
The overall objective of this program of research is to improve sexual health outcomes for women diagnosed with breast or gynecologic cancer. The investigators are developing a multi-component intervention for the four key predictors of sexual health in female cancer survivors: self-image, vaginal symptoms, desire/energy, and relationship-partner concerns. This proposal addresses the evaluation of this last component, relationship-partner concerns. The planned intervention to address these concerns is a psychosexual education partner program (PEPP) delivered by workbook and three follow up phone calls (to coincide with the end of each module) to women and their partners who have experienced a negative change in their relationship since their cancer diagnosis. Ten women with breast or gynecological cancer and their stable partners (ten dyads) will evaluate the content and delivery method of the intervention through self-report questionnaires and a qualitative interview.

ELIGIBILITY:
Eligibility Criteria below apply only to the patient. (The patient's partner must be 18 years of age or older.)

Patient Inclusion Criteria:

1. Age ≥18 female with a history of any stage breast and/or gynecological cancer.
2. Completed primary treatment (chemotherapy, radiation and/or surgery) ≥ 3 months and ≤ 5 years prior to registration.
3. May use concurrent adjuvant endocrine therapy or HER2-targeted therapy while on study.
4. Responds yes to the question "Has there been change in communication and/or intimacy with your partner since your cancer diagnosis?"
5. Ability to read and write English.
6. A stable partner, defined as anyone with whom the woman has had an intimate relationship with for at least 3 months prior to her cancer diagnosis.
7. Both partner and woman must agree to participate in the study and sign informed consent to the study.

Patient Exclusion Criteria:

1. Antidepressants are allowed if a person has been on them for 30 days prior to registration, and dose or treatment is not expected to change.
2. Past history of sexual abuse.
3. Psychiatric disorder such as major depressive disorder, bipolar disorder, obsessive compulsive disorder or schizophrenia. (Defined per medical history and/or patient self-report.)
4. Currently enrolled in another study that addresses sexual health (enrollment in other clinical trials will be allowed).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Attrition rate (feasibility) | Week 6 (+2 weeks)
  After completion of each module the interventionist will contact patients and their partners by phone and document completion of the module's exercise. Anyone who does not provide data both before and after completing the surveys for the study will be considered to be prematurely withdrawn and included in the attrition count. The intervention will be considered feasible if the attrition rate is 25% or less at week 6 (+2 weeks). Withdrawal reasons will be captured and reported by category.

SECONDARY OUTCOMES:
Home practice rate (acceptability) | Week 6 (+2 weeks)
  At each follow up phone call the interventionist will document participant progress and completion of the module's exercise. This documentation will include an assessment of whether or not both participants reviewed the module (yes/no), if no who did not review content, completion of module activities (yes/no), if no which activity was not completed. This documentation will be used to calculate adherence rates by dyad and individual.
Participant experience assessed using Thematic Analysis | Week 6 (+2 weeks)
  Participant experience will be evaluated using the investigator-developed interview guide, which asks questions to assess usefulness, timing, delivery, content and perceived benefit. Research staff will record (either via audio or HIPAA-compliant video platform) participant responses to participant experience questions. Responses will be transcribed and then reviewed by two study team members and discussed in detail. Data analysis will be grounded in the theory of Thematic Analysis, which has been proven to be an effective framework for uncovering meaning in qualitative data. The research team will then connect the codes to try to identify themes for participant experience.
Impact of intervention, measured by Dyadic Sexual Communication (DSC) | Baseline to week 6 (+2 weeks)
  DSC is a single dimensional 13-item scale that measures sexual communication between partners on a Likert scale, 1-disagree strongly to 6- agree strongly. Data will be summarized using descriptive statistics. To measure the effect size, Cohen's d or f, will be calculated for from baseline to week 6.
Impact of intervention, measured by PROMIS® Sexual Function and Satisfaction V2.0 (PROMIS SexF V2) | Baseline to week 6 (+2 weeks)
  PROMIS SexF V2 measures sexual activities, symptoms, functioning, and evaluation of sexual experiences. General screener items ask about sexual activity and reasons for not having sexual activity in the past 30 days. Researchers are encouraged to select the sexual function and satisfaction domains and items that are relevant to the specific sample being studied. For this study, this measure will be administered to both partners. Females will answer the 14 item version and males will answer a 10 item version. In this instrument, higher scores indicate more of the thing being described by the domain. Effect sizes will be calculated from baseline to week 6. Data will be summarized using descriptive statistics. To measure the effect size, Cohen's d or f, will be calculated for from baseline to week 6.
Impact of intervention, measured by Revised Dyadic Adjustment Scale (RDAS) | Baseline to week 6 (+2 weeks)
  RDAS is a 14-item scale with 3 themes (satisfaction, cohesion, and consensus) that measures an individual's perception of the quality of relationship with an intimate partner using a 6 point Likert scale; score range from 0 to 69. Higher scores indicate more positive dyadic adjustment. Scores of 47 and below indicate relationship distress. Data will be summarized using descriptive statistics. To measure the effect size, Cohen's d or f, will be calculated for from baseline to week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Arring, DNP, PhD, RN, OCN, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arring NM, Reese JB, Lafferty C, Barton DL, Carter J. A Sexual Health Self-Management Intervention (Psychosexual Educational Partners Program) for Couples With a History of Breast and Gynecological Cancer: Mixed Methods Feasibility Study. JMIR Form Res. 2025 Oct 21;9:e75743. doi: 10.2196/75743. PMID 41118642